CLINICAL TRIAL: NCT02867748
Title: TVT-ABBREVO Versus SERASIS for the Treatment of Female Urinary Stress Incontinence: 1 Year Outcomes of a Comparative Study With 2 Trans-obturator Sub Mid Urethral Slings
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0141-15-NHR
Record Dates: First submitted 2016-05-08; First posted 2016-08-16 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2017-11

CONDITIONS: Urinary Stress Incontinence
Keywords: tvt abbrevo , Serasis
MeSH Terms: conditions — Urinary Incontinence, Stress

ARMS (2):
- 1 (Experimental): TVT-Abbrevo
  Interventions: Procedure: TVT-Abbrevo
- 2 (Experimental): Serasis
  Interventions: Procedure: Serasis

INTERVENTIONS:
Procedure: TVT-Abbrevo
  Arms: 1
Procedure: Serasis
  Arms: 2

SUMMARY:
Abstract:

Urinary Stress Incontinence (USI)- is a discomforting condition that negatively affects the quality of life of many female individuals and frequently treated by surgical intervention. The incontinence curative operations revolutionized at 1995, with the introduction of the first retro-pubic sub-mid urethral synthetic sling, firstly named Intra-Vaginal Sling-plasty (IVS) and then Tension Free Vaginal Tape (TVT), by Ulmsten and Petros. This was later proposed to be done trans-obturatorly (TOT), for avoiding operative bladder injuries.

Among other peri-operative complications attributed to the commonly used anti-incontinence TOT are the thigh and groin pain. These pains are subjects of concern for patients and physicians worldwide. Another, rare yet very disturbing post-operative complication is erosion of the polypropylene tape into the vagina. TOT palpation at vaginal examination was claimed to be a predictive sign for future erosion of the polypropylene tape into the vaginal cavity.

This current study aims to compare TVT-Abbrevo procedure (12 cm polypropylene tape, Ethicon J&J Somerville, NJ, USA ) to Serasis procedure (softly knitted monofilament non-absorbable polypropylene, Serag-Wiessner, Naila, Germany) for the cure of USI. The purpose of this study is to evaluate the feasibility, the safety and the cure rate of both procedures, as well as documenting the post-operative immediate, and long term thigh and groin pain levels, and dyspareunia. This study is aimed to evaluate the palpability of the implanted tapes at vaginal examination and the possible relation of this to further vaginal tape exposure.

Investigators hypothesized that using Serasis tape, which is made of a softer polypropylene material than rather rigid TVT-Abbrevo polypropylene tape might result in lower pain levels at the short and long term post-operative course, as well as to reduced tape palpability and exposure to the vaginal cavity. investigators believe that favorable results for this study might improve patients' post-operative quality of life and overall satisfaction.

Keywords: Serasis, TVT-Abbrevo, USI, pain, groin, thigh, dyspareunia, safety, urinary stress incontinence, sub mid urethral sling, trans-obturator, TOT, Intra-Vaginal-Sling plasty.

DETAILED DESCRIPTION:
Introduction:

The International Uro-gynecological Association (IUGA) and International Continence Society (ICS) defined urinary stress incontinence (USI) as urine loss condition during effort, physical exertion such as sports activities, or while sneezing or coughing1. USI is not a life threatening condition, yet, if left untreated, it might have a significant negative impact on quality of life of many patients. According to epidemiologic studies woman's age, multi-parity and menopausal status are all risk factors for USI1,2.Treatment options offer changes in life style, and nonsurgical modalities such as pelvic floor muscle training which can be useful in mitigating discomforting symptoms. However, upon failure of conservative treatment, surgery will be recommended for women who are unsuccessful in coping with USI3.

Intravaginal sling-plasty retro-pubic surgical procedure was reported by Ulf Ulmsten and Peter Petrous at 1995 for treating urinary stress incontinence4. Soon after, a study was done on this new procedure now called TVT, which was concluded to be a safe and an efficient ambulatory procedure4-6. This led to a major change with the uro-gynecologic operation preferences, based mainly on the open retro-pubic operations before hands. Trans-obturator sub mid urethral tape procedures (TOT) for treating female urinary stress incontinence were reported then-after, first by Delorme 7, then by De Leval 8. The TOT procedures were designed in order to minimize the incidence of some TVT related adverse effects that might severely impede patient's rehabilitation and health, such as urinary tract injuries, urinary outlet obstruction, bowl penetration and intra-operative bleeding9,10. The TOT procedures' efficacy was claimed to be non-inferior to the TVT, therefore became greatly adopted by uro-gynecologists world-wide9. The fact that the TOT needle passes through the medial compartment of the obturator fossa 2.5-3.0 cm to the obturator vessels and nerves, might explain the incidental post-operative thigh pain10.

Despite the fact that TOT is reported to have low complication rates, there are still complaints on post-operative thigh and groin pain as well as dyspareunia11. Study on a mini TVT, a single incision sling that doesn't pass through the obturator membrane, proved reduced post-operative pelvic and thigh pain, yet many surgeons are reluctant to use mini TVT implants because of reduced cure rates. Dyspareunia, however, occurred with TVT, TOT and mini TVT procedures causing concern with sexually active patients11. Thus TOT procedures are frequently performed and thigh and groin pains are constantly a common complications caused by trans-obturator passage of the sling close to the obturator nerve. The typical TOT post-operative pain is at the thigh, uni or bilateral, yet it was described even at the lumbar spine or hip regions. This might have been due to patient's hips position during operation, but more likely to intra-operative obturator nerve injury or post-operative nerve impact, due to a direct pressure or tape foreign body reaction9. Jean De Leval, Alexandre Thomas and David Waltregny proposed a modified TOT, the TVT-Abbrevo (Ethicon J&J Somerville, NJ, USA). The polypropylene tape's length was reduced to 12 cm. The TVT-Abbrevo was developed in order to avoid extensive tape trans-obturator traumatic passage, reduce amount of mesh in the aponeurotic tissues, and this way to reduce the postoperative pain in the thigh and groin areas9. Their results showed that the group underwent modified TVT-Abbrevo procedure experienced less pain on day 0 than the TVT-Obturator group but not thereafter 9,12. In addition to thigh and groin pain, Sue Ross, in his clinical study was concerned to find that an indicative number of women in TOT group had a palpable polypropylene tape at vaginal examination one year after the surgery13. These findings are rather concerning because risk factors for unfavorable outcomes of tape surgeries are not completely understood. It is hard to state whether palpable tapes will lead to erosions or get absorbed into the vaginal tissue that will result in further complications13,14.

The Serasis (Serag-Wiessner, Naila, Germany) was launched for the potential beneficiary impact of especially soft knitted sling implant on the occurrence and severity of post-operative pain. The ratio behind it is the notion that the tape softness will reduce tissue trauma when the tape is introduced through the obturator plat and maybe less fibrotic tissue reaction as well. There are no comparative studies performed on effectiveness of Serasis tape implantation as an anti-USI procedure, neither a comparison against other polypropylene tapes.

Aims of this study:

In this prospective study investigators wish to aim to compare the Serasis to the TVT-Abbrevo, used for the treatment for USI. Firstly, investigators will evaluate feasibility, the safety and the curative rate of both procedures including the post-operative immediate and long term pain levels as well as the dyspareunia with both groups. Secondly, investigators will evaluate differences in the ability to palpate the Serasis and TVT-Abbrevo tapes at vaginal examination in both groups one year post surgery. In this study investigators focus our attention on rigidity of the Serasis tape versus the common polypropylene tape, which is provided with the TVT-Abbrevo. In addition, investigators will evaluate the significance of previously reported phenomena of vaginal palpability of TVT one year after the implantation 13,14.

Study Hypothesis:

Previous studies showed that the TVT-Abbrevo caused less immediate post-operative thigh and groin pain but was not found in the long term12. This current study hypothesis is that being gently knitted, the Serasis tape, would be superior to the TVT-Abbrevo tape, in terms of post-operative pain levels and severity. Investigators think that Serasis might be an effective solution for the above stated post-operative complications due to its softer monofilament non-absorbable polypropylene tape.

The author presumes that:

1. The objective and subjective curative rates should be around 85% in Serasis group and in TVT-Abbrevo group.
2. Early postoperative pain levels, caused probably by operative trauma, will be the same in Serasis and TVT-Abb groups of patients.
3. The long term post-operative pain levels, dyspareunia and ability to palpate the implanted tape at vaginal examination will be reduced with the Serasis patients' group in comparison to the TVT-Abbrevo groups of patients.

Study significance:

Results of this study will provide important limited information regarding Serasis and TVT-Abbrevo tapes, such as efficacy, immediate and long term post-operative outcomes and vaginal tape palpability and exposure. This data might improve surgeon's decision making and patients' outcome and satisfaction. If adverse clinical postoperative outcomes will be found to be reduced with the gently knitted sling, patient care and quality of life might be improved as well.

Methods:

1. Study design: This is a double arm, prospective and randomized comparative study. Randomization will be done by anesthesiologist flipping a coin right before beginning of the procedure.

The enrolled patients will be given detailed, open and transparent thorough data regarding the study. Patients will sign an informed consent and get randomized onto one of the two study groups, to have either Serasis or TVT-Abbrevo.

The operations will be performed under general anesthesia and the patients will be discharged 8 hours after surgery.

The operations will be performed according with previously medially deviated trans-obturator needle passage11.

Data will be downloaded from the patient's medical charts and collected on interviews by using 3 questionnaires (Pain Q, UDI-6, IIQ-7) and physical exams.

1. Pre-operation: interview+ physical exam+ (Pain Q, UDI-6, IIQ-7).
2. Intra-operative estimate of feasibility and safety: needle passage ease and adjustment (VAS system), estimate blood loss (CC).
3. Before discharge from the hospital: chart data download, interview+ physical exam+ pain questionnaire.
4. Early postoperative follow up: interview and a pain questionnaire by telephone on the 1st post-operative day.
5. 1 month follow up: interview+ physical exam+ Pain Q, UDI-6, IIQ-7 questionnaires, palpability score will be determined at physical exam.
6. 3 months follow up: interview by telephone+ Pain Q, UDI-6, IIQ-7 questionnaires
7. 12 months follow up: interview + Pain Q, UDI-6, IIQ-7 questionnaires, physical exam including objective palpability score determination.

Data will be collected, reviewed and investigated by the researchers. Data collection: 1 year; Data processing: 2 months; Statistical analysis: 2 months; Writing the final thesis: 2 months Duration of the study is planned to be up to 2 years starting in 2015.

2. Subjects:

Inclusion criteria:

Women suffering from urinary incontinence during physical exertion proved by clinical examination.

This study is planned to include 100 patients, 50 women in each group- Serasis and TVT-Abbrevo, based on the assumption of 50% difference in pain levels between the two patient's groups.

The exclusion criterion:

1. Women younger than 30 and older than 80 years old.
2. Women who had surgical procedures involving the pelvic floor, either for the treatment of USI or for Pelvic Organ Prolapse (POP).
3. Women who suffer from advanced POP (POP-Quantification system (POP-Q) stage more than 2).
4. Patients who have absent or incomplete medical records.
5. Women who refuse to participate with the study.
6. Women who are not able to give informed consent or participate with this randomized research study for any other reason.

3. Variables: Demographic data will be collected such as age, background illness, etc.. Preoperative / Intraoperative /Postoperative data collection: medical charts and records, questionnaires on quality of life, urogenital and sexual functioning, surgical procedure that was undertaken, clinical postoperative analysis, pain levels and other intra and post-operative complications will be evaluated using (VAS).

Pain location, severity, onset and duration will be determined at thorough examination by the main researcher. The ability to palpate on the polypropylene tape at vaginal examination will be examined as well (VAS).

The primary outcome measures are the cure or failure of the operation, as well as any adverse effects such as dyspareunia or pain. This will be based upon interview and questionnaires. The second outcome measure is the ability to palpate on the polypropylene tape at vaginal examination.

Statistical methods:

Quantitative data will be presented using mean and standard deviation, median and Ranges, while qualitative data will be presented using frequencies and percentages. Comparison of quantity data between the groups will be examined by comparisons tests: Independent sample t-test or Wilcoxon rank sum test, as appropriate. Qualitative data will be compared among / between groups using Chi square test or Fisher's exact test, as appropriate. Changes over time will be examined. Quantity data will be compared by Repeated measurers, Freidman test, paired sample t-test or Wilcoxon signed ranks test, as appropriate. Ordinal data will be compared by Freidman test or Wilcoxon signed ranks test, and Qualitative data will be compared mainly by McNemar test.

Sample size calculation: for recovering sufficient information investigators will need 100 patients for this study in order to meet the power of 80% with the estimation of 50% difference at pain level.

Estimation of feasibility and safety of the procedures: blood loss (CC), needle passage ease (VAS).

Estimation of pain level at : intercourse, vaginal examination, and of constant pelvic, thigh and groin pain follow up 1 month, 3 months and 12 months after the surgery.(VAS) Estimation of tape palpability: 1 month and 12 months (VAS). Estimation of cure rate: persistent failure, recurrence, or completely dry - Yes/ NO interview.

ELIGIBILITY:
Inclusion Criteria:

* Women suffering from urinary incontinence during physical exertion proved by clinical examination

Exclusion Criteria:

1. Women younger than 30 and older than 80 years old.
2. Women who had surgical procedures involving the pelvic floor, either for the treatment of USI or for Pelvic Organ Prolapse (POP).
3. Women who suffer from advanced POP (POP-Quantification system (POP-Q) stage more than 2).
4. Patients who have absent or incomplete medical records.
5. Women who refuse to participate with the study.
6. Women who are not able to give informed consent or participate with this randomized research study for any other reason

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2016-09; Primary Completion 2018-09 (Actual); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
urinary stress incontinence cure | one year follow up
  Primary outcome measure will be the cure of urinary stress incontinence subjective as reported by the patient in percentage of postoperative residual leak vs preoperative leak.
  Objective cure rate will be the leakage at physical examination cough test with full bladder (200-400ml) verified by US

SECONDARY OUTCOMES:
Safety, intra and postoperative adverse effects | 1 year follow up
  the ability to palpate the sling at vaginal examination (yes/no)

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Western Galilee MC, Nahariya
  - Assuta MC, Tel Aviv

REFERENCES:
- [Background] Citgez S, Onal B, Erdogan S, Demirdag C, Korkmaz M, Demirkesen O, Talat Z, Erozenci A, Cetinel B. Risk Factors for Women to Have Urodynamic Stress Urinary Incontinence at A Turkish Tertiary Referral Center: A Multivariate Analysis Study. Urol J. 2015 Jul 1;12(3):2187-91. PMID 26135936
- [Background] Canel V, Thubert T, Wigniolle I, Fernandez H, Deffieux X. Postoperative groin pain and success rates following transobturator midurethral sling placement: TVT ABBREVO(R) system versus TVT obturator system. Int Urogynecol J. 2015 Oct;26(10):1509-16. doi: 10.1007/s00192-015-2723-8. Epub 2015 May 12. PMID 25963058
- [Background] Ulmsten U, Petros P. Intravaginal slingplasty (IVS): an ambulatory surgical procedure for treatment of female urinary incontinence. Scand J Urol Nephrol. 1995 Mar;29(1):75-82. doi: 10.3109/00365599509180543. PMID 7618052
- [Background] Atan A, Basar MM. A multicenter study of tension-free vaginal tape (TVT) for surgical treatment of stress urinary incontinence. Int Urogynecol J Pelvic Floor Dysfunct. 2000;11(2):130-2. doi: 10.1007/s001920050084. No abstract available. PMID 10805273
- [Background] Nilsson CG, Palva K, Aarnio R, Morcos E, Falconer C. Seventeen years' follow-up of the tension-free vaginal tape procedure for female stress urinary incontinence. Int Urogynecol J. 2013 Aug;24(8):1265-9. doi: 10.1007/s00192-013-2090-2. Epub 2013 Apr 6. PMID 23563892
- [Background] Delorme E. [Transobturator urethral suspension: mini-invasive procedure in the treatment of stress urinary incontinence in women]. Prog Urol. 2001 Dec;11(6):1306-13. French. PMID 11859672
- [Background] de Leval J. Novel surgical technique for the treatment of female stress urinary incontinence: transobturator vaginal tape inside-out. Eur Urol. 2003 Dec;44(6):724-30. doi: 10.1016/j.eururo.2003.09.003. PMID 14644127
- [Background] de Leval J, Thomas A, Waltregny D. The original versus a modified inside-out transobturator procedure: 1-year results of a prospective randomized trial. Int Urogynecol J. 2011 Feb;22(2):145-56. doi: 10.1007/s00192-010-1264-4. Epub 2010 Sep 21. PMID 20857087
- [Background] Menahem N. Tension-free vaginal tape obturator: midterm data on an operative procedure for the cure of female stress urinary incontinence performed on 100 patients. J Minim Invasive Gynecol. 2008 Jan-Feb;15(1):92-6. doi: 10.1016/j.jmig.2007.10.012. PMID 18262152
- [Background] Neuman M, Sosnovski V, Kais M, Ophir E, Bornstein J. Transobturator vs single-incision suburethral mini-slings for treatment of female stress urinary incontinence: early postoperative pain and 3-year follow-up. J Minim Invasive Gynecol. 2011 Nov-Dec;18(6):769-73. doi: 10.1016/j.jmig.2011.08.718. PMID 22024263
- [Background] Tommaselli GA, Formisano C, Di Carlo C, Fabozzi A, Nappi C. Effects of a modified technique for TVT-O positioning on postoperative pain: single-blind randomized study. Int Urogynecol J. 2012 Sep;23(9):1293-9. doi: 10.1007/s00192-012-1758-3. Epub 2012 Apr 18. PMID 22527555
- [Background] Ross S, Robert M, Lier D, Eliasziw M, Jacobs P. Surgical management of stress urinary incontinence in women: safety, effectiveness and cost-utility of trans-obturator tape (TOT) versus tension-free vaginal tape (TVT) five years after a randomized surgical trial. BMC Womens Health. 2011 Jul 22;11:34. doi: 10.1186/1472-6874-11-34. PMID 21781314
- [Background] Ross S, Robert M, Swaby C, Dederer L, Lier D, Tang S, Brasher P, Birch C, Cenaiko D, Mainprize T, Murphy M, Carlson K, Baverstock R, Jacobs P, Williamson T. Transobturator tape compared with tension-free vaginal tape for stress incontinence: a randomized controlled trial. Obstet Gynecol. 2009 Dec;114(6):1287-1294. doi: 10.1097/AOG.0b013e3181c2a151. PMID 19935032
- [Result] Toozs-Hobson P, Freeman R, Barber M, Maher C, Haylen B, Athanasiou S, Swift S, Whitmore K, Ghoniem G, de Ridder D. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for reporting outcomes of surgical procedures for pelvic organ prolapse. Int Urogynecol J. 2012 May;23(5):527-35. doi: 10.1007/s00192-012-1726-y. PMID 22476543
- [Derived] Carter E, Johnson EE, Still M, Al-Assaf AS, Bryant A, Aluko P, Jeffery ST, Nambiar A. Single-incision sling operations for urinary incontinence in women. Cochrane Database Syst Rev. 2023 Oct 27;10(10):CD008709. doi: 10.1002/14651858.CD008709.pub4. PMID 37888839